CLINICAL TRIAL: NCT01649557
Title: A Phase 2, Multicenter, Open-label Study to Assess the Safety and Tolerability of Oral OPC-34712 as Monotherapy in Adult Patients With Schizophrenia
Brief Title: Multicenter, Open-label, Safety and Tolerability Study
Acronym: STEP 210
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-08-210
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-label OPDC-34712 (Experimental)
  Interventions: Drug: OPC-34712

INTERVENTIONS:
Drug: OPC-34712 — oral administered once daily

SUMMARY:
This will be a multicenter, 52 week, open label study to assess the safety and tolerability of oral OPC-34712 (1 to 6 mg) as monotherapy in adult patients with schizophrenia. The study will be conducted on an outpatient basis. Enrollment into the study will be drawn from eligible subjects who have completed participation in Study 331-07- 203 and who, in the investigator's judgment, would benefit from continued treatment with oral OPC-34712.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who participated in 331-07-203 and who, in the opinion of the investigator, have the potential to benefit from continued administration of OPC-34712 for the treatment of schizophrenia.
2. Outpatient status at last visit of Study 331-07-203.

Exclusion Criteria:

1. Sexually active males who are not practicing two different methods of birth control during the study and for 90 days after the last dose of study medication or who will not remain abstinent during the study and for 90 days after the last dose, or sexually active females of childbearing potential who are not practicing two different methods of birth control during the study and for 30 days after the last dose of study medication or who will not remain abstinent during the study and for 30 days after the last dose. If employing birth control, two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pill, birth control depot injection, birth control implant, condom, or sponge with spermicide.
2. Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving open-label OPC-34712.
3. Subjects who during the course of their participation in 331-07-203 were treated in violation of the protocol or who developed ANY exclusion criteria during the course of their participation.
4. Subjects who do not continue to meet all applicable inclusion/exclusion criteria for Protocol 331-07-203 at the last visit (ie, Week 6) of Protocol 331-07-203.
5. Subjects who represent a risk of committing suicide based on an answer of "Yes" to either Question 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) or Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the "Suicidal Ideation" portion of the C-SSRS, or an answer of "Yes" to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory acts or behavior) on the "Suicidal Behavior" portion of the C-SSRS. A subject who has had any suicidal ideation within the last 6 months, any suicidal behaviors within the last two years, or who in the clinical judgment of the investigator presents a serious risk of suicide should be excluded from the study.
6. Subjects who would be likely to require prohibited concomitant therapy during the study.
7. Any subject who, in the opinion of the investigator, should not participate in the study.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (15):
  - Otsuka Investigational Site, Little Rock, Arkansas
  - Otsuka Investigational Site, Escondido, California
  - Otsuka Investigational Site, Garden Grove, California
  - Otsuka Investigational Site, Long Beach, California
  - Otsuka Investigational Site, Oceanside, California
  - Otsuka Investigational Site, Pasadena, California
  - Otsuka Investigational Site, San Diego, California
  - Otsuka Investigational Site, Santa Ana, California
  - Otsuka Investigational Site, Washington D.C., District of Columbia
  - Otsuka Investigational Site, Bradenton, Florida
  - Otsuka Investigational Site, Maitland, Florida
  - Otsuka Investigational Site, St Louis, Missouri
  - Otsuka Investigational Site, Cedarhurst, New York
  - Otsuka Investigational Site, Philadelphia, Pennsylvania
  - Otsuka Investigational Site, Austin, Texas
- Bulgaria (6):
  - Otsuka Investigational Site, Burgas
  - Otsuka Investigational Site, Kazanlak
  - Otsuka Investigational Site, Pazardzhik
  - Otsuka Investigational Site, Plovdiv
  - Otsuka Investigational Site, Radnevo
  - Otsuka Investigational Site, Rousse
- Croatia (2):
  - Otsuka Investigational Site, Rijeka
  - Otsuka Investigational Site, Zagreb
- India (8):
  - Otsuka Investigational Site, Vijaywada, Andh Prad
  - Otsuka Investigational Site, Visakhapatnam, Andh Prad
  - Otsuka Investigational Site, Ahmedabad, Gujarat
  - Otsuka Investigational Site, Bangalore, Karna
  - Otsuka Investigational Site, Mangalore, Karna
  - Otsuka Investigational Site, Pune, Mahara
  - Otsuka Investigational Site, Chennai, Tamil Nadu
  - Otsuka Investigational Site, Varanasi, Uttar Prad
- Philippines (2):
  - Otsuka Investigational Site, Cebu City
  - Otsuka Investigational Site, Mandaluyong
- Romania (4):
  - Otsuka Investigational Site, Arad
  - Otsuka Investigational Site, Bucharest
  - Otsuka Investigational Site, Cluj-Napoca
  - Otsuka Investigational Site, Oradea
- Russia (4):
  - Otsuka Investigational Site, Moscow
  - Otsuka Investigational Site, Moscow Region
  - Otsuka Investigational Site, Saint Petersburg
  - Otsuka Investigational Site, Zagorodnoye
- Serbia (3):
  - Otsuka Investigational Site, Belgrade
  - Otsuka Investigational Site, Kragujevac
  - Otsuka Investigational Site, NoviSad
- Slovakia (5):
  - Otsuka Investigational Site, Bojnice
  - Otsuka Investigational Site, Bratislava
  - Otsuka Investigational Site, Liptovský Mikuláš
  - Otsuka Investigational Site, Rimavská Sobota
  - Otsuka Investigational Site, Žilina
- South Korea (3):
  - Otsuka Investigational Site, Chuncheon
  - Otsuka Investigational Site, Incheon
  - Otsuka Investigational Site, Seoul
- Taiwan (2):
  - Otsuka Investigational Site, Hualien City
  - Otsuka Investigational Site, Taipei
- Ukraine (6):
  - Otsuka Investigational Site, Chernihiv
  - Otsuka Investigational Site, Dnipropetrovsk
  - Otsuka Investigational Site, Kyiv
  - Otsuka Investigational Site, Simferopol
  - Otsuka Investigational Site, Stepanovka
  - Otsuka Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Kane JM, Skuban A, Hobart M, Ouyang J, Weiller E, Weiss C, Correll CU. Overview of short- and long-term tolerability and safety of brexpiprazole in patients with schizophrenia. Schizophr Res. 2016 Jul;174(1-3):93-98. doi: 10.1016/j.schres.2016.04.013. Epub 2016 May 14. PMID 27188270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol was initially approved as a 6-week trial and later extended to a 52-week trial (Amendment 2). The trial enrolled 244 participants at 73 sites in 12 countries. Of the 244 participants, 28 were included in the 52-week enrollment population.
Pre-assignment Details: Trial consisted of a screening visit, treatment phase and safety follow-up at 30 (± 2) days after the last dose of medication. Eligible participants for the trial were those who completed protocol NCT00905307 and who in the investigators judgment would benefit from the treatment.
Groups:
- Prior Brexpiprazole: The participants were grouped based on the medications that they received prior to the trial. The participants in prior brexpiprazole group included the participants who received brexpiprazole prior to the trial. The participants began dosing with brexpiprazole 2 mg daily and the dosage was increased upto 6 mg daily if the dose was well-tolerated.
- Prior Placebo: The participants were grouped based on the medications that they received prior to the trial. The participants in prior placebo group included the participants who received placebo prior to the trial. The participants began dosing with brexpiprazole 2 mg daily and the dosage was increased upto 6 mg daily if the dose was well-tolerated.
- Prior Aripiprazole: The participants were grouped based on the medications that they received prior to the trial. The participants in prior aripiprazole group included the participants who received aripiprazole prior to the trial. The participants began dosing with brexpiprazole 2 mg daily and the dosage was increased upto 6 mg daily if the dose was well-tolerated.
Period: Overall Study
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Started | 179 | 41 | 24
6-week Enrollers | 159 | 35 | 22
52-week Enrollers | 20 | 6 | 2
Completed | 135 | 27 | 15
Not Completed | 44 | 14 | 9
Not completed — Lost to Follow-up | 5 | 0 | 3
Not completed — Adverse Event | 7 | 5 | 1
Not completed — Met withdrawal criteria | 4 | 0 | 0
Not completed — Physician Decision | 8 | 2 | 1
Not completed — Withdrawal by Subject | 15 | 5 | 4
Not completed — Protocol deviation | 0 | 2 | 0
Not completed — Lack of Efficacy | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prior Brexiprazole: The participants were grouped based on the medications that they received prior to the trial. The participants in prior brexpiprazole group included the participants who received brexpiprazole prior to the trial. The participants began dosing with brexpiprazole 2 mg daily and the dosage was increased upto 6 mg daily if the dose was well-tolerated.
- Prior Apripiprazole: The participants were grouped based on the medications that they received prior to the trial. The participants in prior aripiprazole group included the participants who received aripiprazole prior to the trial. The participants began dosing with brexpiprazole 2 mg daily and the dosage was increased upto 6 mg daily if the dose was well-tolerated.
- Total: Total of all reporting groups
Arm/Group | Prior Brexiprazole | Prior Placebo | Prior Apripiprazole | Total
Number analyzed (Participants) | 179 | 41 | 24 | 244
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (10.1) | 41.4 (11.2) | 41.2 (12) | 39.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 17 | 5 | 91
  Male | 110 | 24 | 19 | 153

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) During First 6 Weeks.
Description: AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a participant while enrolled in the trial, whether or not it was considered drug related by the investigator. A serious adverse event (SAE) was any untoward medical occurrence that resulted in death or was life-threatening or required inpatient hospitalization or prolonged hospitalization. A treatment-emergent AE (TEAE) was defined as an AE that started after start of study medication or an AE that continued from baseline and that worsened, was serious, was study medication related, or resulted in death, discontinuation, interruption, or reduction of study medication.
Time Frame: From Baseline up to 6 weeks
Population: The safety dataset comprised of those participants who received at least one dose of open-label brexpiprazole and were enrolled in the 6-week study.
Measure: Number; unit: Participants
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 178 | 41 | 23
Participants
  Participants with AEs | 79 | 19 | 7
  Participants with TEAEs | 78 | 19 | 7
  Participants with serious TEAEs | 4 | 6 | 1
  Participants with severe TEAEs | 2 | 3 | 2

2. Primary Outcome: Number of Participants With AEs in 52-Week Enrollers.
Description: AE was defined as any new medical problem, or exacerbation of an existing problem, experienced by a participant while enrolled in the trial, whether or not it was considered drug related by the investigator. A SAE was any untoward medical occurrence that resulted in death or was life-threatening or required inpatient hospitalization or prolonged hospitalization. A TEAE was defined as an AE that started after start of study medication or an AE that continued from baseline and that worsened, was serious, was study medication related, or resulted in death, discontinuation, interruption, or reduction of study medication.
Time Frame: From Baseline up to 52 weeks
Population: Those participants who received at least one dose of open-label brexpiprazole and who were enrolled in the 52-week study.
Measure: Number; unit: Participants
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 20 | 6 | 2
Participants
  Participants with AEs | 15 | 4 | 2
  Participants with TEAEs | 15 | 4 | 2
  Participants with serious TEAEs | 0 | 0 | 0
  Participants with severe TEAEs | 0 | 1 | 0

3. Secondary Outcome: Change From Baseline in Total Score of Positive and Negative Syndrome Scale (PANSS) by Study Week and at the Last Visit.
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 that indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. The PANSS total score was the sum of the rating scores for 7 positive subscale items, 7 negative subscale items, and 16 general psychopathology subscale items from the PANSS panel. The PANSS total score ranges from 30-210, with higher scores indicating more severe symptoms.
Time Frame: Baseline, Day 4, Week 1, 2, 4, 6, 8, 14, 20, 26, 32, 38, 44, 52 and Last Visit
Population: The efficacy analysis dataset comprised those participants who received study medication of brexpiprazole and had at least one Post-Baseline assessment for PANSS total score.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 178 | 41 | 23
Units on a scale
  Day 4 (N= 169, 36, 22) | 0.11 (5.86) | -1.25 (3.97) | -1.50 (4.97)
  Week 1 (N= 167, 40, 23) | -2.03 (5.49) | -1.53 (7.95) | -1.91 (6.22)
  Week 2 (N= 165, 40, 21) | -2.95 (8.80) | -3.43 (10.68) | -1.86 (6.04)
  Week 4 (N=148, 34, 18) | -4.65 (8.59) | -4.71 (12.85) | -5.39 (6.30)
  Week 6 (N= 138, 31, 15) | -7.51 (8.82) | -7.87 (10.26) | -7.47 (7.22)
  Week 8 (N=20, 6, 2) | -8.80 (8.69) | -5.17 (7.55) | -10.00 (1.41)
  Week 14 (N=20, 6, 2) | -9.85 (8.09) | 6.83 (28.29) | -3.50 (12.02)
  Week 20 (N= 20, 5, 2) | -10.20 (9.12) | -4.60 (10.71) | -6.50 (10.61)
  Week 26 (N= 19, 5, 2) | -12.89 (9.34) | -5.80 (11.56) | -10.50 (7.78)
  Week 32 (N= 18, 5, 2) | -14.67 (10.94) | -3.00 (16.90) | -16.00 (0.00)
  Week 38 (N= 17, 3, 2) | -13.24 (10.97) | -4.67 (10.21) | -13.00 (0.00)
  Week 44 (N= 17, 2, 2) | -16.00 (10.28) | -4.50 (12.02) | -11.50 (2.12)
  Week 52 (N= 16, 2, 2) | -15.00 (10.06) | -5.50 (13.44) | -11.00 (7.07)
  Last visit (N= 176, 41, 23) | -5.99 (11.25) | -2.32 (18.97) | -5.96 (8.27)

4. Secondary Outcome: Change From Baseline in Clinical Global Impression- Severity of Illness Scale (CGI-S) Score.
Description: The severity of illness for each participant were rated using the CGI-S. To perform this assessment, the investigator were to answer the following question: "Considering your total clinical experience with this particular population, how mentally ill was the participant at that time?" Response choices include: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline, Day 4, Week 1, 2, 4, 6, 8, 14, 20, 26, 32, 38, 44, 52 and Last Visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 178 | 41 | 23
Units on a scale
  Day 4 (N= 169, 36, 22) | 0.02 (0.51) | -0.03 (0.29) | 0.05 (0.38)
  Week 1 (N= 167, 40, 23) | -0.08 (0.47) | -0.05 (0.60) | -0.04 (0.37)
  Week 2 (N= 164, 40, 21) | -0.12 (0.63) | -0.18 (0.71) | 0.00 (0.32)
  Week 4 (N= 148, 34, 18) | -0.25 (0.64) | -0.24 (0.82) | -0.22 (0.43)
  Week 6 (N= 139, 31, 15) | -0.40 (0.66) | -0.35 (0.80) | -0.33 (0.49)
  Week 8 (N= 20, 6, 2) | -0.20 (0.77) | 0.17 (0.41) | 0.00 (0.00)
  Week 14 (N= 20, 6, 2) | -0.40 (0.68) | 0.83 (1.60) | 0.50 (0.71)
  Week 20 (N= 20, 5, 2) | -0.55 (0.76) | 0.20 (0.45) | 0.00 (0.00)
  Week 26 (N= 19, 5, 2) | -0.63 (0.90) | 0.00 (0.71) | 0.00 (0.00)
  Week 32 (N= 18, 5, 2) | -0.78 (0.81) | 0.20 (1.10) | -0.50 (0.71)
  Week 38 (N= 17, 3, 2) | -0.71 (0.85) | 0.00 (0.00) | -0.50 (0.71)
  Week 44 (N= 17, 2, 2) | -0.82 (0.81) | 0.00 (0.00) | -0.50 (0.71)
  Week 52 (N= 16, 2, 2) | -0.88 (0.81) | 0.00 (0.00) | -0.50 (0.71)
  Last visit (N= 176, 41, 23) | -0.33 (0.83) | -0.15 (1.20) | -0.30 (0.56)

5. Secondary Outcome: Change From Baseline in Personal and Social Performance Scale (PSP) Total Score.
Description: The PSP was a validated clinician-rated scale that measured personal and social functioning in four domains: socially useful activities (e.g, work and study), personal and social relationships, self-care, and disturbing and aggressive behaviors. Impairment in each of these domains was rated as absent, mild, manifest, marked, severe, or very severe. These ratings were then converted to a total score based on a 100-point scale using algorithms to identify the appropriate 10-point interval, and the rater's judgment that determined the total score within the 10-point interval. Participants with a PSP total score of 71 to 100 were considered to have mild functional difficulty. Scores of 31 to 70 represented manifest disabilities of various degrees and ratings of 1 to 30 indicated minimal functioning that required intense support and/or supervision.
Time Frame: Baseline, Week 1, 2, 6, 26, 52 and Last Visit
Population: as for outcome 3
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 178 | 41 | 23
Units on a scale
  Week 1 (N= 5, 1, 1) | -2.00 (4.82) [-10.00 to 2.00] | -21.00 (0) [-21.00 to -21.00] | -5.00 (0) [-5.00 to -5.00]
  Week 2 (N= 163, 40, 21) | 1.00 (7.11) [-23.00 to 20.00] | 1.50 (8.16) [-13.00 to 30.00] | 0.00 (0.00) [-6.00 to 10.00]
  Week 6 (N= 139, 31, 15) | 5.00 (9.34) [-47.00 to 35.00] | 6.00 (10.86) [-10.00 to 40.00] | 1.00 (5.96) [-8.00 to 16.00]
  Week 26 (N= 19, 5, 2) | 6.00 (5.35) [0.00 to 20.00] | 12.00 (8.07) [-5.00 to 14.00] | 2.50 (3.54) [0.00 to 5.00]
  Week 52 (N= 16, 2, 2) | 13.00 (7.31) [0.00 to 30.00] | 13.00 (1.41) [12.00 to 14.00] | 0.50 (0.71) [0.00 to 1.00]
  Last visit (N= 171, 41, 22) | 4.00 (10.28) [-47.00 to 35.00] | 5.00 (15.10) [-50.00 to 40.00] | 1.00 (5.32) [-8.00 to 16.00]

6. Secondary Outcome: Mean Clinical Global Impression- Improvement Scale (CGI-I) Total Score.
Description: The efficacy of study medication was rated for each participant using the CGI-I. The investigator rated the participants total improvement whether or not it was due to the drug treatment. All responses were compared to the participants condition at Screening/Baseline (i.e, Week 6 visit of Protocol NCT00905307). Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Day 4, Week 1, 2, 4, 6, 8, 14, 20, 26, 32, 38, 44, 52 and Last Visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 178 | 41 | 23
Units on a scale
  Day 4 (N= 169, 36, 22) | 3.70 (0.87) | 3.56 (0.88) | 3.23 (1.15)
  Week 1 (N= 167, 40, 23) | 3.51 (0.89) | 3.73 (0.93) | 3.13 (1.14)
  Week 2 (N= 164, 40, 21) | 3.41 (1.10) | 3.45 (1.28) | 3.38 (1.28)
  Week 4 (N= 148, 34, 18) | 3.14 (1.04) | 3.26 (1.21) | 2.94 (1.21)
  Week 6 (N= 139, 31, 15) | 2.86 (0.99) | 3.03 (1.28) | 2.60 (1.18)
  Week 8 (N= 20, 6, 2) | 2.80 (0.95) | 3.50 (1.22) | 3.00 (1.41)
  Week 14 (N= 20, 6, 2) | 2.75 (0.85) | 3.83 (1.60) | 4.50 (0.71)
  Week 20 (N= 20, 5, 2) | 2.70 (1.03) | 3.20 (1.30) | 4.00 (0.00)
  Week 26 (N= 19, 5, 2) | 2.74 (0.93) | 3.00 (1.41) | 4.00 (0.00)
  Week 32 (N= 18, 5, 2) | 2.56 (0.78) | 3.20 (1.79) | 3.00 (1.41)
  Week 38 (N= 17, 3, 2) | 2.53 (0.87) | 2.67 (1.15) | 3.00 (1.41)
  Week 44 (N= 17, 2, 2) | 2.35 (0.79) | 3.00 (1.41) | 3.00 (1.41)
  Week 52 (N= 16, 2, 2) | 2.31 (0.79) | 3.00 (1.41) | 3.00 (1.41)
  Last visit (N= 176, 41, 23) | 3.04 (1.14) | 3.32 (1.52) | 2.83 (1.19)

7. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Score.
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. In positive subscale, the 7 positive symptom constructs were: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS positive symptom score ranges from 7-49, with higher scores indicating more severe symptoms.
Time Frame: Baseline, Day 4, Week 1, 2, 4, 6, 8, 14, 20, 26, 32, 38, 44, 52 and Last Visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 178 | 41 | 23
Units on a scale
  Day 4 (N= 169, 36, 22) | -0.04 (2.06) | -0.50 (1.36) | 0.09 (2.24)
  Week 1 (N= 167, 40, 23) | -0.66 (1.91) | -0.25 (2.72) | -0.78 (2.76)
  Week 2 (N= 165, 40, 21) | -1.09 (2.92) | -0.70 (3.75) | -0.05 (2.84)
  Week 4 (N= 148, 34, 18) | -1.53 (2.96) | -1.06 (3.95) | -1.11 (2.08)
  Week 6 (N= 138, 31, 15) | -2.36 (3.21) | -2.03 (3.06) | -1.87 (2.39)
  Week 8 (N= 20, 6, 2) | -2.10 (3.02) | -1.67 (2.34) | -2.50 (2.12)
  Week 14 (20, 6, 2) | -2.80 (2.65) | 2.17 (9.04) | 1.00 (4.24)
  Week 20 (20, 5, 2) | -2.60 (3.49) | -1.80 (2.39) | 0.00 (4.24)
  Week 26 (N= 19, 5, 2) | -3.42 (2.99) | -2.60 (2.61) | -3.00 (1.41)
  Week 32 (N= 18, 5, 2) | -3.83 (3.54) | -1.00 (4.85) | -5.00 (1.41)
  Week 38 (N= 17, 3, 2) | -3.71 (4.10) | -2.67 (2.52) | -3.00 (0.00)
  Week 44 (N= 17, 2, 2) | -4.24 (3.53) | -1.50 (2.12) | -4.00 (1.41)
  Week 52 (N= 16, 2, 2) | -3.63 (3.74) | -1.50 (2.12) | -4.50 (3.54)
  Last visit (N= 176, 41, 23) | -1.74 (3.86) | -0.22 (6.04) | -1.43 (2.87)

8. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score.
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. In negative subscale the severity was rated for the following 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS negative symptom score ranges from 7-49, with higher scores indicating more severe symptoms.
Time Frame: Baseline, Day 4, Week 1, 2, 4, 6, 8, 14, 20, 26, 32, 38, 44, 52 and Last Visit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 178 | 41 | 23
Units on a scale
  Day 4 (N= 169, 36, 22) | -0.01 (1.99) | -0.25 (1.00) | -0.86 (2.12)
  Week 1 (N= 167, 40, 23) | -0.47 (2.15) | -0.40 (2.58) | -0.87 (2.44)
  Week 2 (N= 165, 40, 21) | -0.68 (2.61) | -0.83 (2.32) | -1.19 (2.52)
  Week 4 (N= 148, 34, 18) | -1.03 (2.99) | -1.35 (3.02) | -1.94 (2.48)
  Week 6 (N= 138, 31, 15) | -1.70 (3.04) | -1.97 (2.70) | -2.40 (2.61)
  Week 8 (N= 20, 6, 2) | -2.55 (2.68) | -1.00 (2.00) | -1.00 (1.41)
  Week 14 (N= 20, 6, 2) | -2.85 (3.15) | 1.17 (7.05) | -1.50 (2.12)
  Week 20 (N= 20, 5, 2) | -3.00 (3.04) | -0.60 (1.14) | -2.00 (2.83)
  Week 26 (N= 19, 5, 2) | -3.74 (3.43) | -1.20 (1.48) | -2.50 (2.12)
  Week 32 (N= 18, 5, 2) | -4.00 (4.41) | -1.00 (1.87) | -2.50 (3.54)
  Week 38 (N= 17, 3, 2) | -3.94 (3.93) | -0.67 (2.08) | -2.50 (3.54)
  Week 44 (N= 17, 2, 2) | -4.18 (3.61) | -1.00 (2.83) | -2.50 (3.54)
  Week 52 (N= 16, 2, 2) | -4.00 (3.58) | -1.00 (2.83) | -2.00 (1.41)
  Last visit (N= 176, 41, 23) | -1.53 (3.28) | -1.10 (3.85) | -2.09 (2.59)

9. Secondary Outcome: Percentage of Participants With a Positive Response Rate.
Description: Response rate was defined as a reduction of ≥ 30% from Baseline in PANSS total score or CGI-I score of 1 (very much improved) or 2 (much improved) at the Last Visit.
Time Frame: Last Visit
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 179 | 41 | 24
Percentage of participants | 33.5 | 36.6 | 45.8

10. Secondary Outcome: Percentage of Participants Who Discontinued Due to Lack of Efficacy.
Description: Discontinuation rate for the participants discontinued due to lack of efficacy were examined.
Time Frame: Last Visit
Population: as for outcome 3
Measure: Number; unit: Percentage of participants.
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Number analyzed (Participants) | 179 | 41 | 24
Percentage of participants. | 2.8 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: AEs were recorded from Screening (ICF was signed) to Follow-up 30 (± 2) days, up to 52 weeks.
Description: The safety dataset comprised of those participants who received at least one dose of open-label brexpiprazole.
Arm/Group | Prior Brexpiprazole | Prior Placebo | Prior Aripiprazole
Serious Adverse Events (participants affected / at risk) | 4/178 | 6/41 | 1/23
Other Adverse Events (participants affected / at risk) | 31/178 | 10/41 | 4/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prior Brexpiprazole (N=178) | Prior Placebo (N=41) | Prior Aripiprazole (N=23)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Schizophrenia (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Brexpiprazole (N=178) | Prior Placebo (N=41) | Prior Aripiprazole (N=23)
Insomnia (Psychiatric disorders) | 10 | 3 | 0
Extrapyramidal disorder (Nervous system disorders) | 2 | 1 | 2
Headache (Nervous system disorders) | 6 | 5 | 0
Tremor (Nervous system disorders) | 9 | 1 | 0
Anxiety (Psychiatric disorders) | 5 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No